CLINICAL TRIAL: NCT05558813
Title: Prospective Cardiac Magnetic Resonance Imaging Study in Duchenne Muscular Dystrophy (DMD-CMP)
Brief Title: Natural History of Duchenne Muscular Dystrophy Cardiomyopathy (DMD-CMP)
Acronym: DMD-CMP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cancellation of financing by the financier.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP220088; 2020-A03534-35 (Other: ID-RCB Number)
Record Dates: First submitted 2022-04-15; First posted 2022-09-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; dystrophin; cardiomyopathy; cardiac MRI
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DMD-CMP cohort (Experimental): Minor (≥ 6 years) and major patients with genetically proven Duchenne myopathy
  Interventions: Diagnostic Test: Cardiac MRI; Biological: Blood assays

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — two cardiac MRIs with Gadolinum injection at 2-year intervals
Biological: Blood assays — blood samples for the determination of blood biomarkers of heart failure (BNP, NTproBNP) and for the constitution of a biological collection
  Other Names: Blood biobanking

SUMMARY:
The purpose of this study is to describe the progression of tissular and functional myocardial abnormalities in patients with Duchenne muscular dystrophy using cardiac magnetic resonance imaging and blood biomarkers assays.

DETAILED DESCRIPTION:
This study is to describe the progression of tissular (late gadolinium enhancement, T1, T2, ECV assessments) and functional (segmental and global contractility, strain) myocardial abnormalities in patients with Duchenne muscular dystrophy using cardiac magnetic resonance imaging and blood biomarkers assays (troponin I, NTproBNP). Comparison between baseline and 2-years assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria :

* Age >= 6 years
* Genetically proven Duchenne muscular dystrophy
* Affiliation to French medical insurance
* Informed consent provided

Exclusion Criteria :

* Age <6 years
* Left ventricular ejection fraction <30%
* Tracheostomy of hospitalisation for acute respiratory failure <1 year
* Contraindication to MRI: claustrophobia, Gadolinum allergy

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Late gadolinium enhancement burden on cardiac MRI | 2 years

SECONDARY OUTCOMES:
Global T1 on cardiac MRI | 2 years
Global T2 on cardiac MRI | 2 years
Global extracellular volume on cardiac MRI | 2 years
Left ventricular ejection fraction on cardiac MRI | 2 years
Left ventricular systolic circumferentiel strain ejection fraction on cardiac MRI | 2 years
Left ventricular systolic radial strain ejection fraction on cardiac MRI | 2 years
Left ventricular systolic longitudinal strain on cardiac MRI | 2 years
NTproBNP assay in the blood | 2 years
Troponin I assay in the blood | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karim A WAHBI, MD, PhD, Principal Investigator — APHP
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No